CLINICAL TRIAL: NCT07345988
Title: Human Babesiosis in Metropolitan France: a Retrospective and Multicenter Descriptive Analysis.
Brief Title: Human Babesiosis in Metropolitan France
Acronym: BABERETRO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9947
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Human Babesiosis
Keywords: Human Babesiosis
MeSH Terms: conditions — Babesiosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Human babesiosis is a rare zoonosis in Europe caused by protozoa of the genus Babesia, transmitted to humans mainly by ticks of the genus Ixodes. The infection mainly affects individuals who have undergone splenectomy, are immunocompromised, or are elderly, which correspond to the risk factors for the disease. The infection is often underdiagnosed due to its rarity and its often nonspecific clinical presentation (asthenia, fever, flu-like syndrome).

In these high-risk patients in particular, the infection can progress to severe forms, with a mortality rate of up to 20-40%. The clinical picture is then that of a severe infection with multiple organ failure: multifactorial renal failure, respiratory distress due to lesion edema, and disseminated intravascular coagulation. One of the main obstacles to understanding human babesiosis in France and Europe is the low number of cases recorded and published. This situation limits knowledge about the epidemiology of the disease, its clinical presentations, its potential severity, and the effectiveness of the treatments used.

The aim of this study is to describe the epidemiological, clinical, biological, therapeutic, and prognostic characteristics of human babesiosis cases diagnosed in metropolitan France.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥18 years old)
* With a diagnosis of babesiosis confirmed by blood smear or PCR
* Treated in associated centers during the period from January 1, 2000, to December 31, 2024

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with a diagnosis of babesiosis confirmed by blood smear or PCR
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05-04 (Estimated)

PRIMARY OUTCOMES:
Description of the epidemiological, clinical, biological, and therapeutic characteristics of human babesiosis cases diagnosed in mainland France. | Up to 18 months
  This study does not include any evaluation; it simply describes the epidemiological, clinical, biological, and therapeutic characteristics of human babesiosis cases diagnosed in mainland France.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des maladies vectorielles à tiques, CNR Borrelia - CHU de Strasbourg - France, Strasbourg, France